CLINICAL TRIAL: NCT07381920
Title: Effects of Muscle Cooling on Motor Unit Firing of the Quadriceps: A Pilot Feasibility Study
Brief Title: Effects of Muscle Cooling on Motor Unit Firing of the Quadriceps
Acronym: CRYO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Eliott Arroyo, PhD, Assistant Professor, Wake Forest University Health Sciences
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00026267
Record Dates: First submitted 2026-01-19; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: muscle cooling; motor unit behavior; HDsEMG; Quadriceps
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Those randomized to Group A (n=12, 50% men) will perform the thermoneutral condition first, followed by the cooled condition.
  Interventions: Procedure: Cryotherapy
- Sequence B (Experimental): Those randomized to Group B (n=12, 50% men) will perform the cooled condition first, followed by the thermoneutral condition.
  Interventions: Procedure: Cryotherapy

INTERVENTIONS:
Procedure: Cryotherapy — For the cold condition, an Aircast Thigh Pad (Aircast), connected to the Cryo Cuff IC cooler (DJO Global, Vista, California, USA) will be applied to the dominant thigh. The system circulates ice water maintained at approximately 10-15°C with intermittent compression. Cooling duration will be individualized based on mid-thigh skinfold thickness, consistent with published recommendations that account for the effect of subcutaneous tissue on intramuscular cooling9. Participants with a mid-thigh skinfold thickness of 0-10 mm will receive 10 minutes of cooling; those with a skinfold thickness of 11-20 mm will receive 25 minutes of cooling; those with a skinfold thickness of 21-30 mm will receive 40 minutes of cooling; and those with a skinfold thickness of 31-40 mm will receive 60 minutes of cooling. Participants will remain seated for the duration of the cooling treatment.

SUMMARY:
The overall objective of this pilot study is to establish the feasibility and methodological validity of using high-density surface electromyography to characterize motor unit behavior of the quadriceps under thermoneutral and locally cooled conditions, and to generate preliminary data to inform the design of a larger, hypothesis-driven study.

DETAILED DESCRIPTION:
This randomized, cross-over pilot study will recruit 24 healthy young adults (12 men and 12 women) between the ages of 18 and 35 years. Participants will attend two in-person laboratory visits separated by a minimum of 48 hours. Visit 1 will include informed consent, eligibility confirmation, baseline assessments, and familiarization procedures. Visit 2 will include experimental testing under thermoneutral and cooled conditions.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 35 years
* Healthy adults, defined as absence of significant acute/chronic medical condition, injury, and/or illness that may compromise subject safety, limit the ability of the participant to complete the study, and/or compromise the objectives of the study as determined by the Principal Investigator.

Exclusion Criteria:

* Current diagnosis or history of:

  * major metabolic disease (e.g., type I and type II diabetes),
  * neuromuscular disease (e.g., cervical spondylotic radiculomyelopathy, lumbar spondylosis, amyotrophic lateral sclerosis, Guillain-Barré syndrome, and acquired demyelinating polyneuropathies),
  * cardiovascular disease (e.g., stage II hypertension, heart failure, myocardial infarction/ischemia, peripheral vascular disease, Raynaud's phenomenon, or other conditions associated with impaired peripheral circulation),
  * significant myocardial or pericardial diseases (e.g. amyloidosis, constriction),
  * moderate or severe valvular disease,
  * pulmonary/respiratory disease (e.g., asthma, chronic bronchitis, emphysema, chronic obstructive pulmonary disease),
  * cancer,
  * renal disease,
  * liver disease,
  * or anemia.
* Current or recent musculoskeletal injury (e.g. fracture, sprain, dislocation) or any physical disability that precludes safe and adequate testing.
* Pregnancy or breastfeeding.
* Thigh circumference greater than 23 inches
* Mid-thigh skinfold thickness greater 40 mm

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Motor Unit (MU) Yield | Immediately after the intervention
  Number of unique motor units successfully identified (decomposed) from quadriceps HDsEMG recordings during maximal voluntary contractions (MVCs) under thermoneutral and cooled conditions.
HDsEMG Decomposition Accuracy | Immediately after the intervention
  Quality/accuracy of motor unit decomposition from quadriceps HDsEMG recorded during MVCs under thermoneutral and cooled conditions, based on decomposition quality metrics generated by the Delsys Neuromap Precision Decomposition III algorithm.
Proportion of Analyzable MVC Trials | Immediately after the intervention
  Percentage of MVC trials that yield HDsEMG data suitable for motor unit decomposition and analysis under thermoneutral and cooled conditions (successful decomposition and acceptable signal quality).

SECONDARY OUTCOMES:
Slope of MUAP-FR relationship | Immediately after the intervention
  Slope of the linear regression relating MU firing rate to MU action potential amplitude during MVCs under thermoneutral and cooled conditions.
Y-intercept of MUAP-FR relationship | Immediately after the intervention
  Y-intercept of the linear regression relating MU firing rate to MU action potential amplitude during MVCs under thermoneutral and cooled conditions.

OTHER OUTCOMES:
Maximal Voluntary Contraction (MVC) Force | Immediately after the intervention
  Peak knee extensor force (N) achieved during MVC testing under thermoneutral and cooled conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Health and Exercise Science at Wake Forest University, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No